CLINICAL TRIAL: NCT07056075
Title: A Randomized, Controlled, Unblinded Trial Evaluating the Impact of Positive Airway Pressure and Capnometry Compared to Standard Management on the Rate of Desaturations During Nurse-administered Sedation ERCP
Brief Title: Prevention of Desaturations Using Positive Airway Pressure or Capnometry During ERCP
Acronym: PrePAP-ERCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karl Landsteiner University of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Julian Prosenz, Clinician Researcher, Karl Landsteiner University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PrePAP-ERCP
Record Dates: First submitted 2025-06-24; First posted 2025-07-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Desaturation; Hypoxemia; ERCP
Keywords: ERCP; Sedation-related adverse events; desaturation; trial
MeSH Terms: conditions — Hypoxia | interventions — Continuous Positive Airway Pressure; Capnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PAP group (Experimental): Nasal PAP Ventilation System
  Interventions: Device: Nasal PAP Ventilation System
- Control group (Placebo Comparator): Standard management consisting of low-flow oxygen through nasal cannula
  Interventions: Device: Low Flow Oxygen
- Capnometry group (Active Comparator): capnometry and low-flow oxygen through nasal cannula
  Interventions: Device: Low Flow Oxygen; Device: Capnometry

INTERVENTIONS:
Device: Nasal PAP Ventilation System — medical devices that provide nasal positive airway pressure ventilation during endoscopy
  Other Names: nasal positive airway pressure
  Arms: PAP group
Device: Low Flow Oxygen — low flow oxygen though nasal cannula
  Arms: Capnometry group; Control group
Device: Capnometry — capnometry measurement
  Arms: Capnometry group

SUMMARY:
Although sedation during endoscopy is sufficiently safe, desaturations are among the most common side effects of endoscopic retrograde cholangiopancreatography (ERCP) procedures, occurring in approximately 20-30% of cases. Sedation during endoscopy increases the complication rate, and a significant proportion of severe and serious side effects are respiratory/airway-related. However, most patients require sedation to complete the procedure and achieve adequate outcomes during therapeutic ERCP. Therefore, improved measures to increase ERCP safety are needed. Since the demand for anesthesia in many centers already (far) exceeds current capacities, performing additional ERCPs under general anesthesia is not an option. Innovative ways to improve cardiorespiratory monitoring or respiratory management during ERCP could offer a solution without significantly increasing costs. Fortunately, dedicated devices for respiratory management and/or monitoring during endoscopy already exist, but their impact on improving patient safety has not yet been well studied. Therefore, the aim of this prospective, randomized, open-label, non-interventional study is to investigate the effects of non-invasive airway management and respiratory monitoring devices on desaturation rate during endoscopic retrograde cholangiopancreatography.

For this purpose, 288 adult patients (male and female, 18+ years) undergoing ERCP for medical reasons will be enrolled and randomized to one of three groups: (i) airway management using positive airway pressure (PAP group), (ii) additional monitoring using capnography (capnography group), and (iii) a control group with standard monitoring/treatment (i.e., 2 L O2/min via nasal cannula) (control group). Patients are monitored during the ERCP procedure according to medical standards (non-invasive blood oxygen saturation measurement = SpO2, regular non-invasive blood pressure measurement, pulse), and all desaturation events (defined as an SpO2 <85% for any duration according to guidelines) are recorded and treated according to guideline recommendations (the studies do not specify any measures for the (non-)treatment of desaturations). After the procedure, patients are followed (passively) for 30 days (review of medical records) to record late complications. The main outcome parameter is the comparison of the desaturation rate in the PAP versus the control group.

ELIGIBILITY:
Inclusion Criteria:

* undergoing an interventional (intent) ERCP procedure
* 18-99 years
* Male or female
* Nurse-administered sedation

Exclusion Criteria:

* History of allergic reaction to Propofol
* Tracheostomy
* Procedure requiring intubation, general anesthesia, or anesthesiologist backup (acute exacerbation of obstructive lung disease, acute congestive heart failure, supra-glottic or sub-glottic tumor, septic shock, e.g.) according to the endoscopist in charge
* Pregnant patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference in desaturation rate | during endoscopic retrograde cholangio-pancreatography
  Differences of rates of desaturations (i.e., SpO2 <85% for any duration) of the PAP group vs. the standard management group

SECONDARY OUTCOMES:
Difference in desaturation rate | during endoscopic retrograde cholangio-pancreatography
  Differences of rates of desaturations (i.e., SpO2 <85% for any duration) across the three groups
Difference in desaturation rate | during endoscopic retrograde cholangio-pancreatography
  Differences of rates of desaturations (i.e., SpO2 <85% for any duration) of the capnometry group vs. the standard management group
Difference in desaturation rate | during endoscopic retrograde cholangio-pancreatography
  Differences of rates of desaturations (i.e., SpO2 <85% for any duration) of the PAP group vs. the capnometry group
Rates of interventions for hypoxemic events | during endoscopic retrograde cholangio-pancreatography
  Rates of interventions for hypoxemic events in the PAP group vs. the control group
Rates of interventions for hypoxemic events | during endoscopic retrograde cholangio-pancreatography
  Rates of interventions for hypoxemic events in the PAP group vs. the capnometry group
Rates of interventions for hypoxemic events | during endoscopic retrograde cholangio-pancreatography
  Rates of interventions for hypoxemic events in the capnometry group vs. the control group
Lowest SpO2 | during endoscopic retrograde cholangio-pancreatography
  Lowest SpO2 values across the three groups
Median procedure length | during endoscopic retrograde cholangio-pancreatography
  Median procedure length (min) across the three groups
Satisfaction with sedation | Periprocedural
  Endoscopist and patient satisfaction levels concerning the procedure on a Likert scale ("Satisfaction scale" 0-10, 0=worst, 10=best) across the three groups
Rate of sedation-related adverse events | during endoscopic retrograde cholangio-pancreatography
  Rate of sedation-related adverse events across the three groups
Rate of SCOPE | from ERCP up to 30 days after procedure
  Rate of a combined endpoint of serious adverse events and clinical outcomes (SCOPE) across the three groups
  SCOPE (serious adverse events and clinical outcomes in procedural endoscopy) includes:
  30-day all-cause mortality, cardiopulmonary resuscitation1, unplanned intubation or non-invasive ventilation1, single or multiorgan dysfunction due to an endoscopy-related adverse event (AGREE IVa/IVb), rescue or secondary intervention (endoscopic, surgical, or interventional radiology) due to an endoscopy-related adverse event (AGREE IIIa/b), post-ERCP pancreatitis, or target not reached (with necessity of a secondary procedure)
  1 AE occurring after start of the procedure (first dose of sedation administered) until patient leaves recovery room.

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Division of Gastroenterology and Hepatology, Department of Medicine, Medical University Graz, Graz
  - Department of Internal Medicine 2, University Hospital of St Pölten, Sankt Pölten

IPD SHARING:
Plan to Share IPD: No